CLINICAL TRIAL: NCT04804735
Title: Use of Virtual Reality Mask or Music Therapy for Analgesia and Anxiolytic Purpose When Totally Implanted Venous Access Device (IVAD) for Chemotherapy Under Local Anesthesia
Brief Title: Use of Virtual Reality Mask or Music Therapy for Analgesia and Anxiolytic Purpose When Totally IVAD for Chemotherapy Under Local Anesthesia
Acronym: REVCCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Curie (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IC 2020-03
Record Dates: First submitted 2021-03-16; First posted 2021-03-18 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Implanted Venous Access Device
MeSH Terms: interventions — Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- REV : local anesthesia and virtual reality (Experimental): Use of virtual reality device in Implanted Venous Access Device (IVAD) procedure under local anesthesia
  Interventions: Device: REV : local anesthesia and virtual reality
- MUS : local anesthesia and music therapy (Experimental): Use of musicotherapy tool in Implanted Venous Access Device (IVAD) procedure under local anesthesia
  Interventions: Device: MUS : local anesthesia and music therapy
- CONTROL : standard local anesthesia (No Intervention): Implanted Venous Access Device (IVAD) procedure under local anesthesia as standard of care

INTERVENTIONS:
Device: REV : local anesthesia and virtual reality — REV : local anesthesia and virtual reality in Implanted Venous Access Device (IVAD) procedure under local anesthesia
  Arms: REV : local anesthesia and virtual reality
Device: MUS : local anesthesia and music therapy — MUS : local anesthesia and music therapy in Implanted Venous Access Device (IVAD) procedure under local anesthesia
  Arms: MUS : local anesthesia and music therapy

SUMMARY:
Evaluate 2 medical devices on pain average and/or anxiety average in the totally Implanted Venous Access Device (IVAD) procedure under local anesthesia.

DETAILED DESCRIPTION:
Evaluate the efficacy of virtual reality and music therapy on pain average and/or anxiety average in the totally Implanted Venous Access Device (IVAD) procedure under local anesthesia.

ELIGIBILITY:
Inclusion Criteria:

1. Patient aged between 18 and 85 years.
2. Patient with cancer care and having a totally Implanted Venous Access Device (IVAD) procedure under local anesthesia for chemotherapy.
3. Absence of anxiolytic premedication.
4. Patient affiliated to social insurance.
5. Absence of contra-indication to the use of virtual reality, music therapy instrument or local lidocaine anesthesia.
6. Signed informed consent form.

Exclusion Criteria:

1. Patient already participated to this study.
2. Patient deprived of liberty or under legal representative or under curatorship.
3. Psychiatric disease enabling communication.
4. Deafness or visual impairement.
5. Patient under beta-blockers medication.
6. Chronic pain present and not equilibrated before the measured procedure as > 3 by the NRS.
7. Tracheotomy.
8. Low cervical tumor, or bilateral low cervical adenopathies.
9. Compression or jugular stenosis (uni or bilateral).
10. Jugular or subclavian thrombosis.
11. Patient under anticoagulants medication or having hesmostasis troubles.
12. Claustrophobia or thalassophobia inducing the possibility of rejecting the virtual reality mask or music therapy mask.
13. Patients not speaking french.
14. Pregnant and breastfeeding women.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2022-12-06 (Actual); Primary Completion 2023-08-16 (Actual); Study Completion 2023-08-16 (Actual)

PRIMARY OUTCOMES:
mean of pain felt during the whole IVAD procedure | 1 day
  pain means will be measured with the Numerical Rating Scale (NRS) from 0 to 10 with 0 corresponding to no pain and 10 the maximum pain feeling.
mean of anxiety felt during the whole IVAD procedure | 1 day
  Anxiety means will be measured with the Numerical Rating Scale (NRS) from 0 to 10 with 0 corresponding to no anxiety and 10 the maximum anxiety feeling.

SECONDARY OUTCOMES:
Correlation coefficient between the ANI air under the curve and the pain measure with the numerical rating scale. | 1 day
  Correlation coefficient between the ANI air under the curve and the pain measure with the numerical rating scale.
Tolerance evaluated by NRS and responses to the closed questions (dizziness, nausea, suffocating feeling) completed at the end of the procedure. | 1 day
  NRS and responses to the closed questions
Global patient satisfaction of NRS and comparison between the 3 groups. | 1 day
  patient satisfaction of NRS
Pain NRS means felt during the procedure and comparison. | 1 day
  NRS means
Anxiety NRS means felt during the procedure and comparison. | 1 day
  NRS means

CONTACTS AND LOCATIONS:
Overall Officials: Steven LE GOUILL, Pr., Study Director — Institut Curie
Locations (3):
- France (3):
  - Institut Curie, Paris
  - Institut Curie, Saint-Cloud
  - Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: Yes
Sponsor will share de-identified data sets Documents generated under the project will be disseminated in accordance with Institut Curie policies.
Supporting Information: Study Protocol, SAP
Time Frame: Data requests can be submitted starting 9 months after last article publication and will be made accessible for up to 12 months.
Access Criteria: Access to trial individual participant data can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a data sharing agreement (DSA).